CLINICAL TRIAL: NCT02694276
Title: Internet-based Cognitive Behavior Therapy for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate professor, lic. psychologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF pilot ICBT 2015
Record Dates: First submitted 2015-12-14; First posted 2016-02-29 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-based cognitive behavior therapy (Experimental): 10 sessions of ICBT during 10 weeks.
  Interventions: Behavioral: Internet-based cognitive behavior therapy

INTERVENTIONS:
Behavioral: Internet-based cognitive behavior therapy — The CBT treatment lasts for 10 weeks and includes the following: Education on the role of anxiety on cardiac function and the effects of symptom preoccupation and avoidance QoL and depression in AF, creating a vicious cycle; exposure to physical sensations that are similar to AF symptoms (e.g.,palpitations due to physical activity or stress) to reduce fear of these symptoms; exposure to situations or activities previously avoided and abolishment of behaviors that fruitlessly aim to prevent triggering of AF episodes or to control symptoms; and behavioral activation aiming to increase social and physical activity and reduce depressive symptoms. Therapist support is provided at least once weekly through the platform developed for the purpose. Therapists are trained CBT-psychologists.

SUMMARY:
The aim is to evaluate if internet- delivered CBT, based on behavioral activation and exposure principles, improves wellbeing and QoL in symptomatic AF patients.The study will include 30 patients with symptomatic AF despite optimal medical treatment in accordance with current guidelines.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia (irregular heartbeat) affecting 3% of the population. AF is associated with poor quality of life (QoL) and large costs for society. In a considerable proportion of patients, AF symptoms (e.g., palpitations, fatigue, and chest pain) are not alleviated by current medical or interventional treatments. Psychological factors can worsen AF symptoms, and anxiety and depression are common among AF patients. Symptom preoccupation and avoidance of social and physical activities are likely to play important roles in the development of anxiety, depression, disability and healthcare utilization.

The aim is to evaluate if CBT, based on behavioral activation and exposure principles, improves wellbeing and QoL in symptomatic AF patients.

Method: Pilot study with a pre-post-design and no control group. The internet-delivered CBT-program will last for 10 weeks and include weekly therapist support, consisting of online messages and telephone calls.

ELIGIBILITY:
Inclusion Criteria:

A) Paroxysmal AF ≥ once per month that causes moderate to severe symptoms and leads to significant distress or interferes with daily life (i.e. EHRA class ≥ IIb) [31]; B) Age 18-75 years; C) Able to read and write in Swedish.

Exclusion Criteria:

C) Heart failure with severe systolic dysfunction (ejection fraction ≤ 35%); D) Significant valvular disease; E) Other severe medical illness; F) Severe depression or risk of suicide; G) Alcohol dependency. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-12; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in The Atrial Fibrillation Quality of Life (AFEQT) | From baseline to 12 weeks
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction.
Change in The Atrial Fibrillation Quality of Life (AFEQT) | From baseline to 9 months.
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction.

SECONDARY OUTCOMES:
WHODAS 2.0 (12-item version) • | From baseline to 12 weeks.
  Change in general quality of life
WHODAS 2.0 (12-item version) • | From baseline to 9 months.
  Change in general quality of life:
Symptom checklist (SCL) | From baseline to 12 weeks.
  Change in AF related symptoms:
Symptom checklist (SCL) | From baseline to 9 months.
  Change in AF related symptoms:
Atrial Fibrillation Severity Scale | From baseline to 12 weeks.
  Change in symptomatic burden
Atrial Fibrillation Severity Scale | From baseline to 9 months.
  Change in symptomatic burden
Cardiac Anxiety Questionnaire | From baseline to 12 weeks.
  Change in symptom preoccupation:
Cardiac Anxiety Questionnaire | From baseline to 9 months.
  Change in symptom preoccupation
GAD-7 | From baseline to 12 weeks.
  Change in anxiety
GAD-7 | From baseline to 9 months.
  Change in anxiety
PHQ-9 | From baseline to 12 weeks.
  Change in depression:
PHQ-9 | From baseline to 9 months.
  Change in depression
Perceived stress scale | From baseline to 12 weeks.
  Change in stress reactivity
Perceived stress scale | From baseline to 9 months.
  Change in stress reactivity
Change in healthcare consumption and work loss: TIC-P | From baseline to 12 weeks.
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Change in healthcare consumption and work loss: TIC-P | From baseline to 9 months.
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Change in symtomatic burden: Holter ECG. | From baseline to 12 weeks.
  The patient will undergo a 24 h ECG assessment in order to measure objectively symptomatic burden (number and duration of symptomatic AF episodes and symptomatic "non-AF episodes")
Change in symptomatic burden: Holter ECG. | From baseline to 9 months.
  The patient will undergo a 24 h ECG assessment in order to measure objectively symptomatic burden (number and duration of symptomatic AF episodes and symptomatic "non-AF episodes")

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, PhD, Principal Investigator — Karolinska Institutet; Frieder Braunschweig, PhD, Study Director — Karolinska Institutet
Locations (1):
- Department of Clinical Neuroscience, Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Sarnholm J, Skuladottir H, Ruck C, Klaveback S, Olafsdottir E, Pedersen SS, Braunschweig F, Ljotsson B. Internet-Delivered Exposure-Based Therapy for Symptom Preoccupation in Atrial Fibrillation: Uncontrolled Pilot Trial. JMIR Cardio. 2021 Mar 2;5(1):e24524. doi: 10.2196/24524. PMID 33650972